CLINICAL TRIAL: NCT06263725
Title: Protein Restriction (PR) for Weight Loss
Acronym: PR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ALyster
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Diet, Healthy, Body Weight
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restricted dietary protein (Experimental): 5 week intake of a isocaloric diet restricted in protein
  Interventions: Other: Restricted dietary protein; Other: Habitual diet
- Habitul diet (Experimental): 5 week intake of habitual, high protein diet
  Interventions: Other: Restricted dietary protein; Other: Habitual diet

INTERVENTIONS:
Other: Restricted dietary protein — Participants will be allocated to 5 week isocaloric restricted protein intake
Other: Habitual diet — Participants will be follow their habitual, high protein intake

SUMMARY:
Prolonged dietary protein restriction has been shown to increase energy expenditure in mice simultaneously with an increase in plasma FGF21 levels. In overfeeding studies, a protein-restricted diet reduces weight gain in both mice and humans compared with normal and high-protein diets. Further, in energy balance studies, when lean men are provided with a protein-restricted diet for five weeks, an increase in energy intake was necessary to obtain their body weight. However, whether the effect of a protein-restricted diet is the same when consumed by overweight to obese men has divergent results in both mice and humans.

DETAILED DESCRIPTION:
The present study is a randomised intervention study. Inclusion criteria for the study are healthy males age between 25 and 45 years, BMI between 26 and 32, low physical activity level (low aerobic capacity with a VO2 - peak of 30 ± 10 mL/min/kg), non-smoker, not using snuff, not suffering from diabetes, hypertension, or any daily medication use and a high dietary protein intake (≥1,5 g/kg body weight/day). Before the intervention period, the participants complete a two-week run-in period. The run-in period is designed to collect more detailed information about the participant's habitual diet, body weight, and physical activity pattern, as well as habituate the participants in the various tasks they have to complete during the intervention. Then a five-week intervention period is initiated where the participants are randomized to follow one of the following diets for 5 weeks: 1) a diet reduced in protein, replaced by primary carbohydrates (11 E% Protein, 50 E% carbohydrates, 37 E% fat), and 2) a control diet comprising habitual protein content (21E% Protein, 40 E% carbohydrates, 37 E% fat).

In the five-week intervention period, all food and drinks (besides water and coffee) are provided for the participant. All food is weighed to 1 gram of accuracy in meal portions for a seven-day cycle and is delivered to the participant.

During the intervention the volunteers participate in six test days, one every week during the intervention. 48 hours prior to the weekly test, the participants are asked to abstaine from vigorous physical activity. On all the test days, the participants arrive in the morning in a fasted state (no food or drink after 10 pm the night before) by passive transportation.

On the first test day (WT0), body composition is determined by DXA scan, and the total body water content is measured using bioimpedance analysis. Then resting metabolic rate is measured. Still, in the supine position, a blood sample is obtained from an antecubital vein. Biopsies are taken at baseline and at the end of the intervention (WT5). A fat biopsy is obtained from periumbilical subcutaneous adipose tissue and a muscle biopsy from the vastus lateralis muscle. On test day 3, halfway through the intervention, body composition, body water, and resting metabolic rate are measured, and blood is sampled from an antecubital vein. On week tests 1, 2, and 4, resting metabolic rate is measured, and blood sampled. At all visits to the institute, body weight is also measured.

During the intervention the participants wear a Sens motion sensor to monitor daily activity level.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 26 and 32 Low physical activity level Non-smoker Not using snuff Not suffering from diabetes, hypertension, or any daily medication use High protein intake (≥1,5 g/kg body weight/day)

Exclusion Criteria:

-

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Body weight | 5 weeks
  The effect of a prolonged moderate protein-restricted diet on body weight in obese participants.

SECONDARY OUTCOMES:
FGF21 | 5 weeks
  study plasma FGF21 concentrations in relation to energy turnover

CONTACTS AND LOCATIONS:
Overall Officials: Bente Kiens, D.Sci, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Denmark